CLINICAL TRIAL: NCT04067934
Title: The Feasibility of Jumping Based Exercise to Improve Musculoskeletal Outcomes in Children and Adolescents With Inflammatory Bowel Disease (The JUMP IBD Study)
Brief Title: JUMP Inflammatory Bowel Disease Study
Acronym: JUMP IBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN19GA217P
Record Dates: First submitted 2019-07-25; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Paediatrics; Exercise
MeSH Terms: conditions — Inflammatory Bowel Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pilot/feasibility design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jumping exercise (Experimental): High-impact exercise intervention: 3 sessions per week for four weeks Each session will consist of three jumping-based exercises, performed for three sets of various repetitions, following a progressive protocol with increasing volume/intensity.
  Interventions: Behavioral: Jumping Exercise programme

INTERVENTIONS:
Behavioral: Jumping Exercise programme — Four weeks of three jumping-based exercise sessions per week. These sessions will involve basic jumping movements, with approximately 50-100 jumps per session; incorporating 20-30 minutes of exercise.

SUMMARY:
Children and adolescents with inflammatory bowel disease are at increased risk of poor bone and muscle health through a variety of factors, including underlying disease processes, nutritional deficits, and reduced physical activity.

Inflammatory bowel disease can also delay the onset of puberty in children, and pubertal development in adolescents, resulting in sub-optimal adult bone mass, therefore increasing future risk of fractures and osteoporosis. High impact exercise may be a useful additional therapy for adolescents with IBD, as the mechanical strains produced during this type of exercise, through high force muscular contractions and ground reaction forces, can promote bone formation and gains in muscle mass. There have been no previous studies assessing the effects of high impact exercise in IBD, so it is unknown if this type of exercise is feasible in this population. The aim of this study is to assess the feasibility of a short term jumping based exercise intervention for improving muscle and bone outcomes in children and adolescents with inflammatory bowel disease.

DETAILED DESCRIPTION:
This study will incorporate a pilot/feasibility design, aiming to recruit a cohort of 15 inflammatory bowel disease patients of child and adolescent age (10 - 17.9 years). No control group will be recruited.

After potential recruits have contacted the study team to signal their interest in participation, a member of the team will contact them to discuss details of the study in more depth, and assess their suitability for participation against the inclusion/exclusion criteria. If eligible, and willing to participate, they will be asked to attend a baseline session (<28 days prior to exercise intervention) during which they will be afforded the opportunity to ask any questions they may have regarding the study.

This visit will last approximately 1.5 hours. Parent/guardian will also be encouraged to ask any questions they may have. Fully informed written consent with be obtained from the participant's parent/guardian if aged under 16 years, and written informed consent (or assent, depending on competence) will also be taken from the participant. A baseline blood sample will be collected at this session by a research nurse. Participants will complete a range of questionnaires regarding quality of life (IMPACT III, PedsQL Generic Core Scale), fatigue (PedsQL Multidimensional fatigue scale), self-efficacy for exercise. A member of the study team will measure disease activity using a clinical questionnaire (wPCDAI, PUCAI). Demographic and disease history data, and physical measurements including height, sitting height, weight, body composition (bio-electrical impedance) will also be collected. Participants will be provided a wrist-worn accelerometer to measure their habitual physical activity for the proceeding seven days, which they will be instructed to return in a provided pre-paid envelope. A kit will be given for participant to provide a stool sample, to be brought to the following study visit. The exercise intervention will consist of four weeks of three jumping based exercise sessions per week. These sessions will involve basic jumping movements, with approximately 50-100 jumps per session; incorporating 20-30 minutes of exercise. Participants will be requested to attend a one hour face-to-face session at the beginning of each intervention week so a member of the study team can teach them safe and correct execution of each of the prescribed movements for that week. Participants will be provided with an exercise log diary in which they can record adherence to each session, and detail if they have experienced any pain or falls (adverse events), or if anything has prevented them from participating in the prescribed session. Should they be unable to attend any face-to-face session, the exercise diary contains details of the prescribed exercises, and how to perform them. A member of the research team will make telephone contact with research participants and their parent/guardian once per week throughout the four weeks, on any week that they do not attend a face to face exercise session. As a minimum, participants will be expected to attend their first exercise session face-to-face with a member of the research team. Participants will be requested to wear a wrist-worn accelerometer throughout the intervention period, which will be routinely downloaded at each face-to-face session.

Follow-up visits will be completed <14 days post-intervention, at which all of the measurements from the baseline visit will be conducted again (excluding height, habitual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis) at least 6 months prior to study involvement
* aged 10 to 17.9 years (inclusive)
* ability to provide written informed consent, or assent with accompanying parent/guardian consent
* ability to mobilise and perform exercise independently
* disease in remission, or mildly/moderately active, according to weighted Paediatric Crohn's disease activity index (wPCDAI) or Paediatric ulcerative colitis activity index (PUCAI)
* stable medication for >4 weeks prior to study, and no planned changes of medication during study period

Exclusion Criteria:

* lack of capacity to provide consent or assent
* pregnancy (females)
* recent (<12 weeks) surgery, or planned surgery during intervention period
* significant contraindication to high-impact exercise
* significant comorbidity
* use of medication known to affect bone turnover (excluding that used to treat IBD [i.e. glucocorticoids])
* BMI > +3.5 standard deviation score (SDS)
* participating in >2 hours per week structured exercise (excluding school physical education)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise protocol | 4 weeks
  Number of exercise repetitions/sessions completed

SECONDARY OUTCOMES:
Bone metabolism biomarker | Baseline and 4 weeks
  Blood levels of bone alkaline phosphatase
Growth hormone axis | Baseline and 4 weeks
  Blood levels of Growth Hormone (GH)/Insulin-like Growth Factor (IGF) axis
Inflammatory cytokines | Baseline and 4 weeks
  Tumour Necrosis Factor (TNF)-alpha levels
Muscle function | Baseline and 4 weeks
  Jumping mechanography power output
Disease activity | Baseline and 4 weeks
  Faecal calprotectin levels
Health-related quality of life | Baseline, 2 weeks and 4 weeks
  Score on IMPACT III questionnaire: the scale measures disease specific quality of life in paediatric IBD patients; TOTAL Score is measured on a scale of 0 - 100; higher scores indicate better QoL; the questionnaire has Four sub-domains: Well-being, emotional functioning, social functioning and body image; all sub-domains also measured 0 - 100 scale, with higher scores indicating better QoL in that domain
Fatigue | Baseline and 4 weeks
  Score on PedsQL Multidimensional fatigue scale: the scale measures generic fatigue in children and adults; Total score is measured on scale of 0 - 100; higher score indicates less fatigue; three sub-domains - general fatigue, sleep/rest fatigue, cognitive fatigue - scored on same 0 - 100 scale; higher score = less fatigue
Bio-electrical impedance as measure of Body composition | Baseline and 4 weeks
  Bio-electrical impedance

CONTACTS AND LOCATIONS:
Overall Officials: Jarod Sze Choong Wong, MBBS MRCPCH DMedSc, Principal Investigator — University of Glasgow
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No